CLINICAL TRIAL: NCT04668014
Title: The Characteristics and Role of Mucosal Microbiome After Treatment of Clostridioides Difficile Infection
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005228
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sigmoid colon biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research is being done to study the ability of C. difficile to colonize the colonic mucosa of individuals with no prior history of C. difficile infection.

DETAILED DESCRIPTION:
The ability of C. difficile to colonize the mucosa of the colon will be studied in healthy individuals with no history of C. difficile infection who are undergoing colonoscopy for colon cancer/polyp screening purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* No history of C. difficile infection
* Undergoing clinically indicated colonoscopy for colon cancer screening or colon polyp surveillance purposes in the absence of active GI symptoms.

Exclusion Criteria:

* Known active pregnancy
* Other known active gastrointestinal infectious process
* Inflammatory gastrointestinal conditions (microscopic colitis, inflammatory bowel disease, Celiac disease)
* Vulnerable adults
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing screening colonoscopy who have no history of C. difficile infection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Presence of C. difficile within the sigmoid colonic mucosal tissue | 1 day (At time of biopsy)
  C. difficile identified on fluorescence microscopy via FISH staining

CONTACTS AND LOCATIONS:
Overall Officials: Purna Kashyap, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials